CLINICAL TRIAL: NCT04475861
Title: Metabolomics and Wound Healing in Diabetes-Mechanisms and Clinical Value of Arginine Supplement in Patients With Diabetic Foot Ulcers
Brief Title: Metabolomics and Wound Healing in Diabetes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 201702332A3
Record Dates: First submitted 2018-09-18; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2018-06

CONDITIONS: Diabetes Mellitus, Type 2; Infection
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Infections

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-arginine supplements (Experimental): The enrolled subjects will then be randomized into two groups. Study Group: will take a supplementation pill containing 5 g L-arginine (0.5g/ pill, GNC, USA) All the food intake of the subjects during the 4 weeks of the study will be recorded and supervised by responsible dietitians.
  Interventions: Dietary Supplement: L-arginine supplements and nutritional supports
- nutritional supports (No Intervention): The enrolled subjects will then be randomized into two groups. Control group: will take a supplementation pill containing 5 g whey protein (5g/ pack, Santosa,Taiwan).
  All the food intake of the subjects during the 4 weeks of the study will be recorded and supervised by responsible dietitians.

INTERVENTIONS:
Dietary Supplement: L-arginine supplements and nutritional supports — The enrolled subjects will then be randomized into two groups. The subjects will receive either L-arginine (the study group) or another amino acid supplement (the control group), with 60 patients in each group. All the food intake of the subjects during the 4 weeks of the study will be recorded and supervised by responsible dietitians.
  Arms: L-arginine supplements

SUMMARY:
The dysfunction of wound healing in diabetes involves multiple healing processes by diminished inflammatory responses and delayed deposition of matrix components, wound remodeling, and closure. Furthermore, hyperglycemia increases the infection susceptibility of wounds. In Taiwan, we have data demonstrating the nutrition status associated the outcome of diabetic foot ulcer (DFU) acute treatment and value of serum arginine level (in preliminary metabolomics study) to predict one-year healing of DFUs. The arginine has the beneficial effects on wound healing by the action of its metabolites, including vasodilatation, bactericide, growth factors recruitment and collage formation. Nevertheless, its supplement and mechanism in patients with diabetes is still remains unproven. This study aims at (1) defining the effects of arginine supplement, on top of the traditional treatment and risk reduction, on healing outcomes of patients with DFUs, (2) studying the modes of action of arginine supplements in diabetes, and (3) verifying the metabolomics factors and their association with wound healing prospects in patients with DFUs. A total of 120 patients with chronic diabetic foot ulcer will be enrolled and survey in 3 years. Along with standard of care, patients will receive, in a randomized fashion, either arginine (treatment group) or whey protein (control group) 5 g per day supplement for 4 weeks. The wound status will be collected with features in wound size, tissue perfusion, and infection status before and after treatment. Nutritional surveys, nitrogen balance as well as various molecular studies such as metabolomics analysis and neutrophil-to-lymphocyte ratio will be performed to study the association between the molecules of nutrients and the healing

DETAILED DESCRIPTION:
The dysfunction of wound healing in diabetes involves multiple healing processes by diminished inflammatory responses and delayed deposition of matrix components, wound remodeling, and closure. Furthermore, hyperglycemia increases the infection susceptibility of wounds. The wounds noted at distal limb of body, the diabetic foot ulcers, have more significant impacts clinically and socioeconomically compare to those injuries from surgery or pressure sores.

1. Urge for Novel treatments in patients with diabetic foot ulcers:

   1.1. Facts: Diabetic foot ulcer (DFU) is a major complication of diabetes that can lead to limb loss and premature death. According to a report from the International Diabetes Federation in 2017, DFU is also the most common cause of hospitalization for patients with diabetes.

   In Taiwan, 1% of patients with diabetes are admitted to hospital for the treatment of DFU annually. However, considering that the lower-extremity amputation (LEA) rate is around 30%,the treatment outcomes are obviously unsatisfactory.

   1.2. Standard treatment for DFU 1.2.1 In 2016, we formed a Taiwan national working group on diabetic foot under the authorization of Diabetes Association of the Republic of China and subsequently published a Diabetic foot guideline in Taiwan in 2017 (ISBN 978-986-82436-8-2). In addition, I also participated in the writing of a clinical foot care guideline released 2017 by International Diabetes Federation . 1.2.2 These two most updated guidelines detail the diagnosis, management and prevention for patients with DFUs with specifically focused on (1) infection, (2) peripheral artery diseases, (3) wound care and surgical intervention, and (4) off-loading and risks reduction. Suggestions for the appropriate medications for patients with various clinical characteristics were also provided. Nevertheless, in addition to treating acute infections and limb ischemia, the optimum healing of a foot ulcer requires treating the complex biological and molecular events of cell migration and proliferation, and of extracellular matrix deposition, remodeling, and tissue microcirculation. This is why the prognosis for patients with DFU is still unsatisfactory, worldwide. Novel treatments are therefore needed to provide better tissue healing in patients with diabetes. Unfortunately, recent results of well-designed novel treatments for patients with DFU have been disappointing.
2. The role of nutrition in wound healing The relationship between nutrition and wound healing, whether after injury or surgical intervention, has been recognized for centuries and adequate carbohydrate, fat and protein intake is known to be necessary for healing to take place. Wound failure, as reflected by wound infections and/or delayed healing, significantly contributes to the financial burden imposed on health care systems worldwide.

   2.1. Molecular pathogenesis of diabetic wound healing In healthy individuals, the wound healing requires maintenance of multiple signals (cytokines and chemokines) released by keratinocytes, fibroblasts, endothelial cells, macrophages, and platelets. During wound-induced hypoxia, VEGF released by macrophages, fibroblasts, and epithelial cells induces nitric oxide synthase (NOS) resulting in an increase in nitric oxide (NO) levels.

   2.2. Role of nutrition in wound healing in patients with diabetes Studies have shown that changes in energy, carbohydrate, protein, fat, vitamin, and mineral metabolism affect the healing process12. Loss of protein due to protein-calorie malnutrition, the most common form of malnutrition, leads to decreased wound tensile strength, decreased T-cell function, decreased phagocytic activity, and decreased complement and antibody levels,ultimately diminishing the body's ability to defend the wound against infection.

   Furthermore, wounding increases metabolic rates, catecholamine levels, loss of total body water, and cellular protein turnover, resulting in an overall state of catabolism.

   Patients with diabetes have a significantly impaired ability to heal wounds, and therefore, exhibit increased complication rates compared with their euglycemic counterparts. The mechanisms at work are multifactorial and need to be further verified.Recent evidence has shown that patients with diabetes exhibit a diminished early inflammatory response and inhibition of fibroblast and endothelial cell activities. Subsequently, when inflammatory cells eventually arrive at the site of injury, they initiate a prolonged inflammatory phase that results in delayed deposition of matrix components, wound remodeling, and closure. Furthermore, hyperglycemia interferes with the cellular transport of ascorbic acid into fibroblasts and leukocytes and decreases leukocyte chemotaxis. In addition, patients with diabetes are more susceptible to infection2 because of decreased host resistance and phagocytosis ability.
3. Preliminary data highlights the role of L-arginine in wound healing in patients with DFU In our diabetic foot center, we have consistently observed that a lower serum albumin level is an independent risk factor for lower-extremity amputation (LEA) . Furthermore, we identified an association between nutritional status and treatment outcomes in patients with limb-threatening DFU. Using the Mini Nutritional Assessment (MNA) and Geriatric Nutritional Risk Index (GNRI) tools, we confirmed a high prevalence of nutritional problems among these patients. We further identified that the nutritional status of the patients was an independent predictor for acute treatment outcomes.

More recently, we analyzed the effect of metabolomic molecules and clinical and wound characteristics on the 1-year outcomes of wound healing in patients with limb-threatening foot ulcer.

ELIGIBILITY:
Inclusion Criteria:

1. are men or non-pregnant women, aged ≥ 40 years or ≤ 80 years
2. have a history of foot ulcers for more than 1 month
3. have a serum albumin level ≤ 4.0 or an ABI level ≤ 1

Exclusion Criteria:

1. Have active malignancy
2. Have acute gastrointestinal surgery
3. are receiving dialysis
4. have heart failure (NYHA Fc ≥ 3), liver cirrhosis (Child class > B), or myocardial infarction in the past 3 months,
5. have wounds complicated with persistent osteomyelitis or Charcot deformity
6. are receiving hydroxyurea or steroid treatment
7. have alcohol abuse, any mental or physiological condition that may interfere with dietary intake, and those who are unable to follow orders or cooperate.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10-31 (Estimated); Primary Completion 2018-12-01 (Estimated); Study Completion 2025-06-18 (Estimated)

PRIMARY OUTCOMES:
PEDIS | up to 1 months
  Wound assessment was recorded using the PEDIS system

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided